CLINICAL TRIAL: NCT00533663
Title: Healing Touch During Chemotherapy Infusions for Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IRB-07696; BRSADJ0007 (Other: OnCore)
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Touch; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Care + Healing Touch (HT) (Experimental): A a gentle, non-invasive form of energy-balancing work that promotes relaxation and can help manage the side effects of chemotherapy. It occurs every other week (during their infusion).
  Interventions: Procedure: Healing Touch; Other: Standard care
- Standard Care + Guided relaxation (Active Comparator): Guided relaxation every other week (during their infusion).
  Interventions: Other: Standard care; Procedure: guided relaxation
- standard care only (Active Comparator): Standard care
  Interventions: Other: Standard care

INTERVENTIONS:
Procedure: Healing Touch — every other week (during their infusion)
  Arms: Standard Care + Healing Touch (HT)
Other: Standard care — Adriamycin, cyclophosphamide, and paclitaxel administered as standard of care
Procedure: guided relaxation
  Arms: Standard Care + Guided relaxation

SUMMARY:
To study if Healing Touch is effective during chemotherapy treatment for breast cancer

DETAILED DESCRIPTION:
To study the effectiveness of Healing Touch provided during chemotherapy infusions on the experience of women undergoing treatment for breast cancer. Healing Touch (HT) is a gentle, non-invasive form of energy-balancing work that promotes relaxation and can help manage the side effects of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:- Stage I or II breast cancer

* Post-operative
* Concurrent enrollment on a treatment protocol of 8 weeks of adriamycin + cyclophosphamide given every other week followed by 8 weeks of paclitaxel given every other week
* ECOG Performance Status: 0 to 2
* Speak and read English

Exclusion Criteria:- Previous chemotherapy exposure

- Concomitant energy-work interventions (HT, Reiki, QiGong, acupuncture).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
FACT-B summary score | Baseline, 6 wks, 14 wks

SECONDARY OUTCOMES:
Domain scores for FACT-B; BSI-18; FACIT-Fatigue; nausea measured on a Likert scale | Baseline, 6 wks, 14 wks

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Turner, RN, NP, Principal Investigator — Stanford University; Alice "Ellie" Guardino, RN, NP, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States